CLINICAL TRIAL: NCT00595283
Title: Early Intervention in Depression: Dyadic Emotion Development Therapy for Preschool Children
Brief Title: Effectiveness of Parent-Child Interaction and Emotion Development Therapy in Treating Preschool Children With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joan Luby, MD, Principal Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH080163 (NIH); R34MH080163 (NIH); DSIR 84-CTS
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Depression
Keywords: Preschool Onset Major Depressive Disorder; Preschool Depression; Emotion Development; Parent Child Interaction
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants assigned to Parent-Child Interaction Therapy-Emotional Development
  Interventions: Behavioral: Parent Child Interaction Therapy-Emotion Development (PCIT-ED)
- 2 (Active Comparator): Participants assigned to Developmental Education Parenting Intervention
  Interventions: Behavioral: Developmental Education Parenting Intervention (DEPI)

INTERVENTIONS:
Behavioral: Parent Child Interaction Therapy-Emotion Development (PCIT-ED) — PCIT-ED includes fourteen 1-hour therapy sessions over 14 weeks. Sessions will focus on positive parent-child interactions skills, ways to manage emotions, and relaxation techniques.
  Other Names: PCIT-ED
  Arms: 1
Behavioral: Developmental Education Parenting Intervention (DEPI) — DEPI includes 14 weekly, 1-hour education sessions covering a range of child development and parenting topics. Classes are in a small group format and will emphasize emotional and social development.
  Other Names: DEPI
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of parent-child interaction therapy that includes an emotion development component in treating depression in preschool children.

DETAILED DESCRIPTION:
While growing up, children experience a range of emotions that change with development and environment. Although all young children experience sadness at times, a main characteristic of young children is their ability to experience joy and excitement in pleasurable childhood activities. When a child seems perpetually sad and no longer seems interested in previously enjoyed activities, the child may be showing signs of early onset depression. Children who are depressed are at increased risk for a wide range of social, psychological, physical, and achievement-related problems. Two previous studies have established the validity of early onset depressive syndrome in preschoolers, confirming the need for treatment during the preschool period. This study will specifically adapt parent child interaction therapy (PCIT), a proven effective treatment for preschool disruptive disorders, for use in preschoolers with depression and will include an additional component to focus on emotion development (ED). The study will evaluate the effectiveness of PCIT-ED in treating depression in preschool children.

Participation in this two-stage study will last 16 weeks and will consist of initial assessments, 14 weeks of therapy, and a final assessment. Stage I will be used to assess the acceptability and reliability of the PCIT-ED manual, which will guide the treatment sessions. The protocol and assessment schedule will be the same for Stage I participants and Stage II participants assigned to PCIT-ED.

The initial assessments will include both child and parent participants. Child participants will be asked to complete a series of tasks, which will include playing with games and toys, making selections based on feelings, completing stories started by a research assistant, and participating in other activities designed to be fun and exciting. Parents will be interviewed about their child's feelings, emotions, behaviors, and development and also about how their child gets along at home, in school, and with friends. Parents will also answer questions concerning their own mental health and drug history, parenting style, and moods.

Participants will then be randomly assigned to receive PCIT-ED or Developmental Education Parenting Intervention (DEPI). Participants in both groups will attend fourteen 1-hour therapy sessions over a period of 14 weeks. For those assigned to PCIT-ED, most sessions will include both parent and child participants, but some will include parents only. During the parent-only sessions, the goals and procedures of upcoming therapy visits will be explained to parents. During sessions with both parent and child, participants will be taught positive parent-child interaction skills, ways to manage emotions, and relaxation techniques. After each therapy session, participants will be given homework that will involve practicing the skills learned in therapy sessions at home. At three points during the study, parents will also be asked to complete a brief questionnaire about their thoughts and feelings toward the therapy process. The therapy sessions for the participants assigned to DEPI will provide basic education in all areas of preschool development, with emphasis on social and emotional development. The initial assessments will be repeated for all participants at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV symptom criteria for MDD based on parent report on PAPA
* Currently resides and has resided with primary caregiver for more than 6 months prior to study entry

Exclusion Criteria:

* Neurologic disorder (e.g., seizure disorder, closed head injury)
* Autistic spectrum disorder
* Has an IQ of less than 70, based on past testing or clear marked developmental delay
* Currently participating in psychotherapy
* If taking a psychotropic medication, must remain on stable dose of that medication throughout the course of study participation

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Depression diagnosis and severity using the Preschool-Age Psychiatric Assessment (PAPA) for major depressive disorder (MDD) module | Measured at Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Joan L. Luby, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine Early Emotional Development Program, St Louis, Missouri, United States

REFERENCES:
- [Derived] Hennefield L, Whalen DJ, Wood G, Chavarria MC, Luby JL. Changing Conceptions of Death as a Function of Depression Status, Suicidal Ideation, and Media Exposure in Early Childhood. J Am Acad Child Adolesc Psychiatry. 2019 Mar;58(3):339-349. doi: 10.1016/j.jaac.2018.07.909. Epub 2019 Jan 8. PMID 30768413